CLINICAL TRIAL: NCT03448328
Title: Influence of Pea Protein Supplementation on Recovery From Exercise-induced Muscle Damage
Brief Title: Pea Protein Supplementation and Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Roquette Freres (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0165
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Muscular Injury
Keywords: muscular strength; inflammation; protein
MeSH Terms: conditions — Inflammation | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pea Protein (Experimental): NUTRALYS pea protein supplement
  Interventions: Dietary Supplement: NUTRALYS pea protein supplement
- Whey Protein (Experimental): Whey protein supplement
  Interventions: Dietary Supplement: Whey Protein
- Apple juice (Active Comparator): Apple juice
  Interventions: Dietary Supplement: Apple juice

INTERVENTIONS:
Dietary Supplement: NUTRALYS pea protein supplement — 0.3 grams of protein per kilogram of body weight before and after eccentric exercise, and each of 4 mornings of recovery
  Arms: Pea Protein
Dietary Supplement: Whey Protein — 0.3 grams of protein per kilogram of body weight before and after eccentric exercise, and each of 4 mornings of recovery
  Arms: Whey Protein
Dietary Supplement: Apple juice — 1.2 calories per kilogram body weight before and after eccentric exercise, and each of 4 mornings of recovery
  Arms: Apple juice

SUMMARY:
The purpose of this study is to determine if supplementation with NUTRALYS pea protein isolate compared to whey protein and apple juice (carbohydrate, non-protein control) before, during, and after a 90-minute bout of eccentric exercise can attenuate exercise-induced muscle damage, inflammation, and delayed onset of muscle soreness (DOMS), and speed recovery of muscle function.

DETAILED DESCRIPTION:
Study participants will be randomized to the NUTRALYS pea protein supplement, whey protein, or apple juice (parallel group design). Study participants will come to the lab at 7:00 am Monday through Friday in an overnight fasted state and provide a blood sample (maximum of 30 ml or two tablespoons). The blood samples will be analyzed for various measures of muscle damage and inflammation, and extra samples will be stored for additional measurements depending on funding.

After the blood draw, participants will provide a muscle soreness rating. Next, the two protein sources (pea and whey protein), will be consumed at a weight adjusted amount (0.3 grams of protein per kilogram of body weight), and administered under double blind procedures. The amount of apple juice will be adjusted to body weight (1.2 calories per kilogram body weight).

Four muscle function tests will be conducted: vertical jump, bench press, leg-back strength, and anaerobic power through the 30-second Wingate test. These performance tests will be administered before and after the 90-minute eccentric muscle exercise bout, and each of the following four mornings of recovery.

After taking the four performance tests, participants will engage in 90-minutes of eccentric exercise. Immediately following exercise, participants will provide a muscle soreness rating and a blood sample, ingest another protein dose (0.3 g/kg) (or apple juice), and then take the four muscle function tests. Participants will return at 7 am in an overnight fasted state four days in a row after the eccentric exercise bout, and provide muscle soreness ratings and blood samples followed by ingestion of the protein supplements or apple juice. Following ingestion of the supplements, participants will take the four muscle function tests.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, 18 to 55 years of age.
* Non-athlete, and not engaged in regular resistance training (less than 3 sessions per week).
* BMI under 30 (non-obese).
* At "low risk" status for cardiovascular disease (as determined with a screening questionnaire).
* Agree to avoid the use of protein and large-dose vitamin/mineral supplements (above 100% of recommended dietary allowances), herbs, and all medications (in particular, NSAIDs such as ibuprofen and aspirin) during the week of the project.

Exclusion Criteria:

* Inability to comply with study requirements.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current, active history of coronary heart disease, stroke, cancer, diabetes, rheumatoid arthritis, high blood pressure, kidney disease, liver disease, blood disease, hormonal disease, or metabolic disease.
* History of cancer in the 5 years prior to the screening visit (except skin or cervical cancer that was successfully treated).
* Current use of any type of medication (or unwillingness to stop use of over-the-counter medications two weeks before the start of the study).
* Recent history of musculoskeletal trauma (fracture, strain, sprain, etc.) that has not fully healed prior to baseline testing.
* Females: pregnant or breastfeeding; or body weight under 100 pounds.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Serum Creatine kinase | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle damage marker

SECONDARY OUTCOMES:
Serum Myoglobin | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle damage marker
Serum Lactate Dehydrogenase | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle damage marker
Delayed onset of muscle soreness | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Self-reported perception of muscle soreness, 1-10 scale
Vertical jump | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle performance, vertical jump height
Bench press | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle performance, bench press to exhaustion with weighted bar (75% body weight for men, 50% for women)
Leg-back strength | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Muscle performance, leg-back strength with a dynamometer
30-second Wingate cycle test | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Anaerobic power cycling test, peak and average anaerobic power
Serum C-reactive protein | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  Inflammation measurement
Plasma cytokine panel | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after)
  IL-6, IL-8, IL-10, MCP-1, IL-1ra, GCSF

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Depends on the journal where the paper will be published.